CLINICAL TRIAL: NCT02978768
Title: The Effect of the Practice of Tai Chi 6-Form Sports Apparatus and Mental Training on Cognition, Self Care, Mood and General Health in Patients With Mild and Moderate Alzheimer's Disease: a Prospective Study.
Brief Title: Tai Chi 6-Form Sports Apparatus With Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Alice May-Kuen Wong, Attending Physician, Chang Gung Memorial Hospital
Allocation: Non-Randomized | Model: Factorial | Masking: None
Other Study IDs: 99-3780B
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Alzheimer Disease
Keywords: dementia; Tai Chi; mental training; cognitive rehabilitation
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Exercise (Experimental): First year, the investigators investigate the effect of 12-week Tai Chi 6-Form accompanied with music rhythm for patients with mild and moderate AD in behavioral and general health, functional and cognitive decline.
  Interventions: Other: Exercise
- Cognitive training (Experimental): Second year, the investigators investigate the effect of 12-week computer-based cognitive training games for patients with mild and moderate AD in behavioral and general health, functional and cognitive decline.
  Interventions: Device: Computer-based cognitive training
- Physico-Mental training (Experimental): Third year, the investigators investigate the effect of 12-week Physico-Mental rehabilitation Wii (PM Wii) for patients with mild and moderate AD in behavioral and general health, functional and cognitive decline.
  Interventions: Device: Physico-Mental rehabilitation Wii

INTERVENTIONS:
Other: Exercise — First year, the investigators investigate the effect of 12-week Tai Chi 6-Form accompanied with music rhythm for patients with mild and moderate AD in behavioral and general health, functional and cognitive decline.
  Arms: Exercise
Device: Computer-based cognitive training — Second year, the investigators investigate the effect of 12-week computer-based cognitive training games for patients with mild and moderate AD in behavioral and general health, functional and cognitive decline.
  Arms: Cognitive training
Device: Physico-Mental rehabilitation Wii — Third year, the investigators investigate the effect of 12-week Physico-Mental rehabilitation Wii (PM Wii) for patients with mild and moderate AD in behavioral and general health, functional and cognitive decline.
  Arms: Physico-Mental training

SUMMARY:
The objective of the present project is to develop complementary and alternative medicine (CAM) for The Chang Gung Dementia Center to alleviate the symptoms and signs of patients with Alzheimer Disease, an approach aiming at decreasing the burden on family, society and nation.

DETAILED DESCRIPTION:
According to statistics in Taiwan, two to four percent the elderly of aged more than 65 years old have dementia. As the decreasing birth rate and the advancement of medical care making life expectancy getting longer, the society in Taiwan is aging with a fast pace, leading to a tremendous increase of patients suffering dementia. Many studies have shown that Tai Chi Chuan can improve quality of life, cardiopulmonary function, pain control, mentality, endurance, flexibility, balance, can decrease the possibility of incidental, and enhance immunity and sleep quality in the elderly. Many studies showed that higher physical activity or mental training is associated with reduced risk for Alzheimer Disease. However, Tai Chi Chuan could be a little difficult for elderly people with dementia because they can't remember so that the investigators have designed Tai Chi 6-Form sports apparatus and the clinical trial was done for health and stroke elderly people. Also, the investigators have developed a mental training program for patients with Alzheimer Disease. The objective of the present project is to develop complementary and alternative medicine (CAM) for The Chang Gung Dementia Center to alleviate the symptoms and signs of patients with Alzheimer Disease, an approach aiming at decreasing the burden on family, society and nation.

1. Study aims during the first year: the investigators investigate the effect of Tai Chi 6-Form accompanied with music rhythm for patients with dementia to remember in behavioral and general health, functional and cognitive decline as well as family caregiver's satisfaction, the use of health care services, and recommendation for other people among patients with mild and moderate Alzheimer Disease.
2. Study aims during the second year: the investigators investigate the effect of mental training with computer mind training games on behavioral and general health, functional and cognitive decline as well as the use of health care services and family caregiver's satisfaction and recom mendation for other people among patients with mild and moderate Alzheimer Disease.
3. Study aims during the third year: the investigators investigate the effect of tele-Tai Chi 6-Form and mental training on line which are to combine to physico-mental rehabilitation Wii (PM Wii) on behavioral and general health, functional and cognitive decline as well as the use of health care services and family caregiver's satisfaction and recommendation for other people among patients with mild and moderate Alzheimer Disease. According to Tai Chi 6-Form, the investigators will develop the software to watch Tai Chi 6-Form exercise on computer on line. The patient can copy Tai Chi 6-Form movement accompanied with previous music rhythm at home. Therefore, Tai Chi 6-Form and mental training which are a great benefit to patients with dementia will be popular at home or in the community. Patients with dementia return back to the community.

ELIGIBILITY:
Inclusion Criteria:

* Mild and Moderate Alzheimer's Disease(AD) participants.

Exclusion Criteria:

* Pacemaker patients.

Ages: 59 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Balance | Up to 3 year
  Outcome measures showed that mild and moderate AD participants received 12-week Tai Chi 6-Form exercise training can improved at balance score, and 12-week computer-based cognitive training may be able to improve their ability to understand instructions and reflected in task execution. In this study, 12-week PM Wii shows no significant difference at balance performance or cognitive function, probably due to the insufficient training intensity and lack of sensory feedback. However, tele-care system is the development trends in the future undoubtedly.

CONTACTS AND LOCATIONS:
Overall Officials: Alice M Wong, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No